CLINICAL TRIAL: NCT02394808
Title: 2-week Dispensing Cross-Over Evaluation of Marketed Silicone Hydrogel Contact Lenses in an Indian Population
Brief Title: 2-week Evaluation of Marketed Silicone Hydrogel Contact Lenses in Indian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5625
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2017-03

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Lens 1 (Experimental): senofilcon A (Approved contact lens material)
  Interventions: Device: senofilcon A; Device: lotrafilcon B
- Test Lens 2 (Active Comparator): lotrafilcon B (Approved contact lens material)
  Interventions: Device: senofilcon A; Device: lotrafilcon B

INTERVENTIONS:
Device: senofilcon A — One fresh pair of contact lenses worn for 11 (+/-2) days, for a minimum of 6 hours per day
Device: lotrafilcon B — One fresh pair of contact lenses worn for 11 (+/-2) days, for a minimum of 6 hours per day

SUMMARY:
The primary objective of this study is to evaluate the clinical performance of two marketed silicone hydrogel contact lenses in an Indian population in the following areas: physiological characteristics, comfort characteristics and vision characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand English, and sign the Statement of Informed Consent and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be 18 and less than 40 years of age.
4. The subject's corrected spherical equivalent distance refraction must be in the range of -1.00 to -5.00D in each eye with visual acuity of 20/25 provided study lenses in each eye.
5. The subject must have less than -1.00 D of cylindrical refraction.
6. The subject must have best corrected visual acuity of 20/25 or better in each eye.
7. The subject must be an adapted soft contact lens wearer in both eyes.
8. The subject must have normal eyes.

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued)
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia.
5. Any previous, or planned ocular or interocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.).
6. Any grade 3 or greater slit lamp findings (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g. past peripheral ulcer, or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
7. Any ocular infections
8. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
9. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment
10. History of binocular vision abnormality or strabismus.
11. Any infectious disease (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV) by self report.
12. Employee of the investigational clinic (e.g. investigator, Coordinator, Technician)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chennai, Tamil Nadu, India

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 54 subjects were enrolled in this study. Of the enrolled subjects all 54 were dispensed a study lens. Of the dispensed 52 completed the study while 2 were discontinued.
Groups:
- Senofilcon A/ Lotrafilcon B: Subjects randomized to this sequence first wore the senofilcon A lens and then wore the lotrafilcon B lens.
- Lotrafilcon B/Senofilcon A: Subjects randomized to this sequence first wore the lotrafilcon B lens and then wore the senofilcon A lens.
Period: Period 1
Arm/Group | Senofilcon A/ Lotrafilcon B | Lotrafilcon B/Senofilcon A
Started | 25 | 29
Completed | 25 | 28
Not Completed | 0 | 1
Not completed — Unsatisfactory lens fitting | 0 | 1
Period: Period 2
Arm/Group | Senofilcon A/ Lotrafilcon B | Lotrafilcon B/Senofilcon A
Started | 25 | 28
Completed | 24 | 28
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least one study lens.
Groups:
- Dispensed Subjects: All subjects that were dispensed at least one study lens throughout the duration of the study.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.83 (4.621)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 54
Region of Enrollment [Number; unit: participants]
  India | 54

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Comfort
Description: Subjective Overall Comfort was evaluated using the Contact Lens User Experience Comfort scores (CLUE). CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: 11 days Post fit
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Senofilcon A: Subjects that wore the senofilcon A lens in either the first or second period of the study.
- Lotrafilcon B: Subjects that wore the lotrafilcon B lens in either the first or second period of the study.
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 48 | 48
units on a scale | 58.65 (18.685) | 59.44 (16.458)

2. Primary Outcome: Subjective Overall Quality of Vision
Description: Subjective Overall quality of Vision was evaluated using the Contact Lens User Experience Comfort scores (CLUE). CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: 11 days post fit
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 48 | 48
units on a scale | 55.60 (16.490) | 58.71 (14.035)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1 month per subject.
Arm/Group | Senofilcon A | Lotrafilcon B
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days